CLINICAL TRIAL: NCT04527939
Title: Results of the Comparative Analysis of Invasion Depth of Extraperitoneal Rectal Neoplasms Between Three-dimensional Endorectal Ultrasonography and Magnification Chromoendoscopy
Brief Title: Analysis of Extraperitoneal Rectal Neoplasms Between 3D Endorectal Ultrasonography and Magnification Chromoendoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Alfonso Bustamante, Principal Investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9076079
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Rectal Cancer; Rectal Cancer Stage I
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Extraperitoneal rectal cancer stage 1
Who Masked: Investigator
Masking Description: Only investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three-dimensional endorectal ultrasonography (Active Comparator): three-dimensional endorectal ultrasonography
  Interventions: Procedure: three-dimensional endorectal ultrasonography
- magnification chromoendoscopy. (Sham Comparator): magnification chromoendoscopy.
  Interventions: Procedure: three-dimensional endorectal ultrasonography

INTERVENTIONS:
Procedure: three-dimensional endorectal ultrasonography — three-dimensional endorectal ultrasonography

SUMMARY:
ERUS-3D and CMI demonstrated good diagnostic accuracy in parietal staging of rectal extraperitoneal neoplasms, however with greater efficiency of the endoscopic method. The association of studies can improve diagnostic efficacy and influence the most appropriate approach.

DETAILED DESCRIPTION:
Larger lesions present less chance of deep parietal invasion. The methods show moderate agreement with each other for lesion size and distance from the anal verge and good agreement for the rectal wall percentage of involvement. Circumferential or almost circumferential lesions have a greater chance of postoperative stenosis. Patients with more advanced lesions on AP who underwent radical resections had lower overall survival.

ELIGIBILITY:
Inclusion Criteria: patients with diagnosis of mid or distal rectum neoplasms stage 1 -

Exclusion Criteria: advanced rectal cancer (stage II, III or IV)

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2023-08-07 (Estimated)

PRIMARY OUTCOMES:
Degree of parietal invasion (T), | immediately after the procedure
  Patients with Stage T after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine School, Sao Paulo University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
comparative analysis of invasion depth of extraperitoneal rectal neoplasms between three-dimensional endorectal ultrasonography and magnification chromoendoscopy.

REFERENCES:
- [Result] Nahas SC, Nahas CSR, Bustamante-Lopez LA, Pinto RA, Marques CFS, Cecconello I. Outcomes of surgical treatment for patients with distal rectal cancer: A retrospective review from a single university hospital. Rev Gastroenterol Mex (Engl Ed). 2020 Apr-Jun;85(2):180-189. doi: 10.1016/j.rgmx.2019.05.009. Epub 2020 Feb 11. English, Spanish. PMID 32057523
- [Result] Kawaguti FS, Franco MC, Martins BC, Segateli V, Marques CFS, Nahas CSR, Pinto RA, Safatle-Ribeiro AV, Ribeiro-Junior U, Nahas SC, Maluf-Filho F. Role of Magnification Chromoendoscopy in the Management of Colorectal Neoplastic Lesions Suspicious for Submucosal Invasion. Dis Colon Rectum. 2019 Apr;62(4):422-428. doi: 10.1097/DCR.0000000000001343. PMID 30730457
- [Result] Pinto RA, Correa Neto IJ, Nahas SC, Rizkalah Nahas CS, Sparapan Marques CF, Ribeiro Junior U, Kawaguti FS, Cecconello I. Efficacy of 3-Dimensional Endorectal Ultrasound for Staging Early Extraperitoneal Rectal Neoplasms. Dis Colon Rectum. 2017 May;60(5):488-496. doi: 10.1097/DCR.0000000000000781. PMID 28383448